CLINICAL TRIAL: NCT06673576
Title: Assessment of The Accuracy of Complete Crown 3D Superimposition Technique Relative to The Gold Standard Technique for Digital Quantification of Volumetric Soft Tissue Changes in The Esthetic Zone
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: British University In Egypt (Other)
Collaborators: Cairo University (Other)
Responsible Party: Principal Investigator, Ahmed Mohamed Hassan, Assistant Lecturer, Cairo University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 131024
Record Dates: First submitted 2024-10-13; First posted 2024-11-05 (Actual); Last update posted 2024-11-05 (Actual); Status verified 2024-11

CONDITIONS: Volume Assessment; Gummy Smile

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Patients assigned for esthetic crown leghthening (Experimental)
  Interventions: Diagnostic Test: Complete crown technique for superimposition; Diagnostic Test: Gold standard technique for superimposition

INTERVENTIONS:
Diagnostic Test: Complete crown technique for superimposition — the complete crown technique, the crown of the tooth corresponding to the gingival margin under evaluation will be selected using the paint method and circular selection tool. The same selection process will be applied to the moving model.
Diagnostic Test: Gold standard technique for superimposition — the gold standard technique, adjacent intact teeth and a portion of the palatal gingiva will be selected. Superimpositions will be executed utilizing the software's iterative closest point algorithm (ICP).

SUMMARY:
The aim of this study is to assess the precision of the complete crown technique employed for the superimposition of 3D models, specifically in the quantitative volumetric evaluation of gingival tissues. This technique was initially introduced in an in-vitro study by Dritsas et al. (2023) as a means to achieve an accurate, reproducible, and simple method for quantification of gingival recession.

This study will involve the analysis of digital models in. ply format acquired through intraoral scanning of patients scheduled for esthetic crown lengthening, with predefined inclusion and exclusion

DETAILED DESCRIPTION:
A digital model T0 (presurgical scan) will be acquired, and the mesh structure will undergo meticulous examination to identify any instances of voids or distorted mesh networks.

Patients will be followed-up for 6 months then undergo the second intraoral scan T6 (6 months follow-up). The resultant mesh structure will be carefully inspected for any defects.

The digital models in. ply format corresponding to T0 (presurgical scan) and T6 (6 months follow-up) will be imported into the BlenderForDental5 software. Notably, the T6 model will be imported twice. Each model will go through a trimming process utilizing the arch cut tool. Subsequently, a base will be created for each model employing the model base tool. A thorough inspection is performed to identify any potential voids in the model base. In cases where voids are detected, the "fill holes" tool will be employed to rectify and fill any voids present within the model base.

Utilizing the superimposition tool, an initial manual alignment of the digital models will be performed, followed by the superimposition procedure. The T0 model will be designated as the reference model, while the first T6 model will be chosen as the moving model. The second T6 model will be designated as the moving.001 model. For the complete crown technique, the crown of the tooth corresponding to the gingival margin under evaluation will be selected using the paint method and circular selection tool. The same selection process will be applied to the moving model. In the case of the gold standard technique, adjacent intact teeth and a portion of the palatal gingiva will be selected. Superimpositions will be executed utilizing the software's iterative closest point algorithm (ICP). A heat map will be generated to verify the accuracy of the superimposition process.

Models will be exported in superimposed orientations to the Geomagic software for the measurement of superimposition accuracy, specifically the root mean square of the tooth corresponding to the gingival margin where volumetric changes are of interest, using the 3D compare tool in Geomagic software.

ELIGIBILITY:
Inclusion Criteria:

1. Patients requiring esthetic crown lengthening.
2. Full-mouth plaque and bleeding score not exceeding 20%.
3. Presence of at least 2.5 mm keratinized tissue width (Pontoriero & Carnevale, 2001).
4. Patients showing motivation to comply with post-operative care instructions and follow-up appointments.

Exclusion Criteria:

* 1. Systemic health conditions that contraindicate or affect healing of periodontal surgery.

  2. Patients requiring prosthetic crowns or restorations in the esthetic zone. 3. Gummy smile with normal tooth proportions. 4. Patients treated with medications known to affect the gingiva (Phenytoin, Cyclosporine and Nifedipine).

  5. Smokers. 6. Pregnant and nursing females.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 12 (Estimated)
Dates: Start 2024-03-15 (Actual); Primary Completion 2025-02-15 (Estimated); Study Completion 2025-05-15 (Estimated)

PRIMARY OUTCOMES:
Superimposition accuracy | 6 months
  Models will be exported in superimposed orientations to the Geomagic software for the measurement of superimposition accuracy, specifically the root mean square of the tooth corresponding to the gingival margin where volumetric changes are of interest, using the 3D compare tool in Geomagic software.

SECONDARY OUTCOMES:
Marginal and Volumetric changes | 6 months
  For assessing changes at the gingival margin level, all three models will be selected, and a crosssection will be generated at the center of the targeted tooth, followed by linear measurements.
  To evaluate volumetric changes, a Boolean modifier will be applied between the T0 model and the T6 model. Excess mesh vertices will then be removed using the clean model tool. Subsequently, the excised gingival margin will become readily apparent and quantifiable, allowing for the measurement of its volume through the utilization of the 3D print module within the BlenderForDental software.

CONTACTS AND LOCATIONS:
Locations (1):
- Cairo University, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: Yes